CLINICAL TRIAL: NCT05513781
Title: Investigation of Factors Causing Knee Hyperextension During Walking in Chronic Stroke Patients by Electromyographic Method
Brief Title: Investigation of Factors Causing Knee Hyperextension During Walking in Chronic Stroke Patients
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Atılım University (Other)
Responsible Party: Principal Investigator, Suleyman Korkusuz, Principal Investigator, Hacettepe University
Other Study IDs: E-59394181-604.01.02-39134
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Stroke
Keywords: Gait Analysis; Stroke; Knee Hyperextension; Electromyography
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic stroke patients with knee hyperextension

SUMMARY:
In this study, it is aimed to examine the factors that cause knee hyperextension in chronic stroke patients. Although the presence of weakness or spasticity in the quadriceps muscle, weakness or spasticity in the plantar flexors, and weakness of the dorsiflexors, hamstrings and gastrocnemius muscle are shown in the literature as the cause of hyperextension of the affected knee in hemiplegic patients, there is a comprehensive study that shows the effect of both muscle strength and spasticity in the lower extremity muscles. there are no studies.

The hypotheses of the study are:

Hypothesis 1:

H0: There is no relationship between knee hyperextension in the stance phase of gait and lower extremity muscle strength in stroke patients.

H1: There is a relationship between knee hyperextension in the stance phase of gait and lower extremity muscle strength in stroke patients.

Hypothesis 2; H0: There is no relationship between knee hyperextension in the stance phase of gait and lower extremity spasticity in stroke patients.

H1: There is a relationship between knee hyperextension in the stance phase of gait and lower extremity spasticity in stroke patients.

Hypothesis 3; H0: There is no relationship between knee hyperextension and electromyographic muscle activations in chronic stroke patients.

H1: There is a relationship between knee hyperextension and electromyographic muscle activations in chronic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 40-65
* At least 6 months have passed since the stroke
* Ambulation with or without a walking aid (walker, cane, or tripod)
* Being between 0-3 points according to the Modified Rankin Score
* Getting a score of 24 or higher on the Mini Mental Test
* Presence of hyperextension in the stance phase of gait
* Volunteering to participate in the study

Exclusion Criteria:

* Having a history of more than one stroke
* Known presence of dementia
* Having a known orthopedic, psychiatric or other neurological disease
* Having a situation that prevents communication
* Having a history of surgery involving lower extremities and gait

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Stroke Patients with Knee Hyperextension
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Movement Analysis | Baseline
  Reflective signs will be placed at certain anatomical points of the participants. Participants will be asked to walk a distance of 5 meters. The three-dimensional positions of these reflective marks will be recorded with the 8-camera Vicon motion capture system. Then it will be examined in computer environment using Blade software.
Electromyographic Measurements | Baseline
  Electromyography (EMG) is frequently used in the literature for motion analysis evaluations. It shows the amplitude of the electrical activity of the muscles. In this study, 8-channel Delsys Bagnoli desktop cable electromyography system (Delsys (Delsys Inc., USA)) will be used. EMG; It shows whether the muscles are active during movement, when they are active and how active they are. In this study, the muscles to be measured by EMG: tibialis anterior, medial gastrocnemius, medial hamstrings, rectus femoris, gluteus medius and the lower part of the latismus dorsi are planned.

SECONDARY OUTCOMES:
Muscle Strength Evaluation | Baseline
  Manual muscle testing will be performed on patients' hip flexors, hip extensors, hip abductors, hip adductors, knee flexors, knee extensors, dorsiflexors, and plantar flexors. A score between 0 and 5 will be given according to the manual muscle test, the ability of the muscles to move against gravity in certain positions, and the resistance of the movement against gravity.
Spasticity Evaluation | Baseline
  The spasticity of the lower extremity muscles (quadriceps, hip extensors, hip adductors, hip internal retractors and plantar flexors) will be evaluated according to the Modified Ashworth Scale. The spasticity assessment will be scored between 0 and 4 according to the resistance of the muscles to passive movement.

CONTACTS AND LOCATIONS:
Overall Officials: Kadriye Armutlu, Prof. Dr., Study Chair — Hacettepe University; Süleyman Korkusuz, MSc, Principal Investigator — Hacettepe University; Sibel Kibar, Assoc. Prof., Study Chair — Atılım University; Serdar Arıtan, Asst.Prof, Study Chair — Hacettepe University; Nihat Özgören, MSc, Study Chair — Hacettepe University; Ali Naim Ceren, Msc, Study Chair — Hacettepe University; Büşra Seçkinoğulları, MSc, Study Chair — Hacettepe University; Ayla Fil Balkan, Assoc.Prof, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Altındağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moseley A, Wales A, Herbert R, Schurr K, Moore S. Observation and analysis of hemiplegic gait: stance phase. Aust J Physiother. 1993;39(4):259-67. doi: 10.1016/S0004-9514(14)60486-4. PMID 25026421
- [Background] Roth EJ, Merbitz C, Mroczek K, Dugan SA, Suh WW. Hemiplegic gait. Relationships between walking speed and other temporal parameters. Am J Phys Med Rehabil. 1997 Mar-Apr;76(2):128-33. doi: 10.1097/00002060-199703000-00008. PMID 9129519
- [Background] Cooper A, Alghamdi GA, Alghamdi MA, Altowaijri A, Richardson S. The relationship of lower limb muscle strength and knee joint hyperextension during the stance phase of gait in hemiparetic stroke patients. Physiother Res Int. 2012 Sep;17(3):150-6. doi: 10.1002/pri.528. Epub 2011 Dec 7. PMID 22147298